CLINICAL TRIAL: NCT01502592
Title: A Pilot Study of Pre-Operative, Single-Dose Ipilimumab and/or Cryoablation in Early Stage/Resectable Breast Cancer
Brief Title: Pre-Operative, Single-Dose Ipilimumab and/or Cryoablation in Early Stage/Resectable Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-202
Record Dates: First submitted 2011-12-29; First posted 2011-12-30 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer; Invasive Adenocarcinoma of the Breast
Keywords: MDX-010 (Ipilimumab); Cryoablation; Total mastectomy planned; 11-202
MeSH Terms: conditions — Breast Neoplasms | interventions — Cryosurgery; Ipilimumab

ARMS (3):
- Cryoablation alone (Experimental): This is a pilot study evaluating the safety and tolerability of pre-operative, single-dose ipilimumab and/or cryoablation in patients with early stage/resectable breast cancer.
  Interventions: Procedure: Cryoablation
- Ipilimumab alone (Experimental): This is a pilot study evaluating the safety and tolerability of pre-operative, single-dose ipilimumab and/or cryoablation in patients with early stage/resectable breast cancer.
  Interventions: Biological: Ipilimumab
- Ipilimumab & Cryoablation (Experimental): This is a pilot study evaluating the safety and tolerability of pre-operative, single-dose ipilimumab and/or cryoablation in patients with early stage/resectable breast cancer.
  Interventions: Procedure: Cryoablation; Biological: Ipilimumab

INTERVENTIONS:
Procedure: Cryoablation — OncCore Biopsy (+ Cryo) Date*
  * Pre- and post- cryo MRI
  * Core biopsy x ≥3
  * Cryoablation Optional pre-surgery MRI day prior or day of Mastectomy Date* Safety assessment 30 (+/-10) days after surgery research bloods 30 (+/-10) days after surgery.*
  Arms: Cryoablation alone; Ipilimumab & Cryoablation
Biological: Ipilimumab — Ipilimumab Appt. with Med Onc Ipilimumab administered Core Biopsy Date*
  * MRI
  * Core biopsy x ≥3 Optional pre-surgery MRI biopsy prior or day of Mastectomy Date* Safety assessment 2-3 weeks post-mastectomy (co-ordinated with off-study surgery follow-up appt if feasible) and then every 2-3 weeks thereafter until at least 12 weeks post ipilimumab date. # Research bloods 30 (+/-10) days after surgery.
  Arms: Ipilimumab & Cryoablation; Ipilimumab alone

SUMMARY:
This study is being done to evaluate the safety of two strategies called "cryoablation" and "immune therapy" in women with curable early stage breast cancer. "Cryoablation" is a procedure performed by an expert doctor called a radiologist. The radiologist uses (magnetic resonance imaging (MRI) to insert a needle directly into a cancer. Very cold temperatures are then applied through the needle to kill the cancer cells. Some of the killed cancer cells will be broken into pieces that can be recognized by a person's immune system.

The "immune therapy" in this study is a drug called ipilimumab. Normally the immune system makes "T cells" that can kill cancer cells when turned on. The cancer-killing T cell activity is controlled by a molecule called CTLA4. Ipilimumab works by turning off CTLA4. Turning off CTLA4 allows the cancer-fighting T cells to remain active Ipilimumab is an antibody drug has been made in a laboratory for patient use and was recently approved by the United States Food and Drug Administration (FDA) for the treatment of patients with a type of skin cancer called melanoma. An antibody is a normal protein that the immune system uses to find and kill germs like bacteria and viruses. This study is being done because the researchers believe that when cryoablation is combined with immune therapy, a person's immune system can be trained to recognize that person's cancer. This may prevent that cancer from coming back in the future. In other words, it is hoped that by adding cryoablation with ipilimumab before the mastectomy, the body will remain cancer free long after the mastectomy is performed. The first step in determining whether cryoablation and immune therapy can be used to cure breast cancer is to evaluate the safety of each strategy alone and then in combination in a small group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 years or older
* Confirmed histologic diagnosis of invasive adenocarcinoma of the breast, including MSKCC pathology confirmation
* ER, PR and HER2 testing in progress(i.e. on outside or MSKCC biopsy report)
* HER2-positive pathology is permitted
* Operable tumor measuring ≥1.5 cm in maximal diameter
* Any nodal status
* Multifocal and multicentric disease is permitted.
* Synchronous bilateral invasive breast cancer is permitted
* No indication of distant metastases
* Total mastectomy planned
* Tumor amenable to cryoablation as determined by radiologist
* ECOG performance status score of 0 or 1

Screening laboratory values must meet the following criteria:

* White blood cells (WBCs) ≥ 2000/μL
* Absolute neutrophil count (ANC) ≥ 1500/μL
* Platelets ≥ 100 x 103/μL
* Hemoglobin ≥ 11.0 g/dL
* Serum creatinine ≤ 2 mg/dL (or glomerular filtration rate ≥ 40 ml/min)
* AST ≤ 2.5 x upper limit of normal (ULN)
* ALT ≤ 2.5 x ULN
* Bilirubin within normal limits (except subjects with Gilbert's syndrome, who must have total bilirubin < 3.0 mg/dL)
* Negative HIV screening test
* Negative screening tests for Hepatitis B and Hepatitis C.
* Patients with positive results that do not indicate true active or chronic infection may enroll after discussion and consensus agreement by the treating physician and principal investigator.
* Women of childbearing potential (WOCBP) must be using an acceptable method of contraception to avoid pregnancy throughout the study and for at least 3 months after the last dose of ipilimumab in such a manner that the risk of pregnancy is minimized. See below for the definition of WOCBP.
* WOCBP must have a negative serum pregnancy test within 14 days of the first study intervention.
* Women must not be breastfeeding.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.
* Definition of WOCBP
* Women of childbearing potential include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal. Post menopause is defined as:
* Amenorrhea ≥ 12 consecutive months without another cause and a documented serum follicle stimulating hormone (FSH) level >35 mIU/mL
* Women with irregular menstrual periods and a documented FSH level > 35 mIU/mL
* Women on hormone replacement therapy (HRT) Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential.

Exclusion Criteria:

* Inflammatory breast cancer
* Medical history and concurrent diseases
* Autoimmune disease: subjects with a documented history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease are excluded from this study as are subjects with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]). Subjects with motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome) are excluded from this study.
* Any underlying medical or psychiatric condition, which in the opinion of the investigator, will make the administration of study drug hazardous or obscure the interpretation of AEs, such as a condition associated with frequent or poorly controlled diarrhea.
* Prohibited Treatments and/or Therapies

  a) Chronic use of immunosuppressants and/or systemic corticosteroids (used in the management of cancer or non-cancer-related illnesses). However, use of corticosteroids is allowed for the treatment of immune related Adverse Events (irAEs), or adrenal insufficiency.
* Any non-oncology vaccine therapy used for prevention of infectious diseases within 4 weeks prior to first dose of ipilimumab.
* Prior treatment with a CD137 agonist, ipilimumab or other CTLA4 inhibitor;
* Prior investigational agents within 4 weeks prior to first dose of ipilimumab;
* Prior therapy with any anti-cancer agents including chemotherapy, adjuvant chemotherapy, immunosuppressive agents, surgery or radiotherapy within 4 weeks prior to first dose of ipilimumab.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
safety | 1 year
  of pre-operative ipilimumab administration and intratumoral cryoablation administered either alone or in combination in patients with early stage breast cancer. Safety will be evaluated for all treated subjects using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events v4.0 (CTCAE).
tolerability | 1 year
  If 5 of the 6 patients in study arm A and 5 of the 6 patients in study arm B are without an AE necessitating delay in surgery, we will enroll 6 additional patients into study arm C. If 5 or 6 of these 6 patients in study arm C are without an AE necessitating delay in surgery, the regimen will be considered safe/tolerable for further study. Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events v4.0 (CTCAE).

SECONDARY OUTCOMES:
Efficacy | 1 year
  exploratory correlative studies will be performed to evaluate anti-tumor and immunological response pre- and post-treatment in individuals. Comparisons with other study participants will also be conducted. Breast cancer tissue specimens, axillary lymph nodes specimens where available, and peripheral blood samples will be studied.

CONTACTS AND LOCATIONS:
Overall Officials: Heather McArthur, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/